CLINICAL TRIAL: NCT05866016
Title: Effectiveness of Modular Skilled Birth Attendant Training to Improve the Competencies of Service Providers and Maternal Newborn Health in Nepal: A Randomized Control Pilot Trial
Brief Title: Effect of Skill Birth Attendant Training to Improve the Competency of Service Providers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health Gandaki Province, Nepal (Other Government)
Collaborators: Ministry of Health and Population, Nepal (Other Government); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Gandaki_MNHstudy_2022_2025
Record Dates: First submitted 2023-05-01; First posted 2023-05-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Competencies of Midwives; Cost-benefit Analysis of Modular Training

STUDY DESIGN:
Intervention Model Description: The competencies of skilled birth attendants who receive modular training will be compared with those of skilled birth attendants who receive existing standard training.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The outcomes assessor and care provider will be masked to minimize the biases. Trainers will be outcomes assessors and trainees who complete modular training and provide maternal and child health services are considered as care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skill birth attendants who trained on new modular training package (Experimental): Maternal and child health service providers (skilled birth attendants) will be trained using modular training that covers both theory and practical sessions on midwifery skills.
  Auxiliary nurse midwives should complete modules 1, 2, and 3 whereas nurses will get modules 1, 2, 3, and 4.
  The training will be implemented in National Health Training Center-accredited training sites/ hospitals.
  Interventions: Behavioral: Skill birth attendant training
- Skill birth attendants who trained on existing standard training package (Active Comparator): Maternal and child health service providers (auxiliary nurse midwives and nurses) get training based on the existing standard skilled birth attendant training curriculum of Nepal. This is a two-month-long integrated skill birth attendant package implemented in National Health Training Center-accredited training sites.
  The midwifery competencies of these service providers will be assessed and compared with the competencies of experimental groups.
  Interventions: Behavioral: Skill birth attendant training

INTERVENTIONS:
Behavioral: Skill birth attendant training — It is an intervention targeted to enhance the competencies of Maternal Neonatal Health (MNH) service providers (skilled birth attendants) in Nepal. It is a capacity-building intervention that is expected to contribute to reducing maternal and neonatal morbidities and mortalities by improving the midwifery competencies (knowledge, attitudes, and skills) of MNH service providers.

SUMMARY:
This clinical trial's primary goal is to compare birth attendants' competencies. It aims to answer the questions:

* Does the new modular training package enhance the competencies of skilled birth attendants?
* Does the competencies of skilled birth attendants relates to improving maternal and neonatal health outcomes in Nepal?
* Is this training module a cost-effective intervention?

Participants' knowledge, attitude, and skills will be assessed and it will be compared with standard training groups: Researchers will compare the competencies of birth attendants who receive modular training versus standard training to see if an increment in competencies is associated with maternal and neonatal health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Health workers should be Auxiliary Nurse Midwives and Nurses working in birthing centers where at least 10 birth managed in the last year
* Health workers (Auxiliary Nurse Midwives and Nurses) who are committed to providing maternal and neonatal health services and priority for permanent service holders.
* Who passes at least the first module (Online module) to participate in modular training

Exclusion Criteria:

* Health workers (Auxiliary Nurse Midwives ad Nurses) who do not provide maternal and neonatal health service
* Health workers other than Auxiliary Nurse Midwives and Nurses though they provide maternal neonatal health services in government health facilities
* Health workers working in private health facilities

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness assessment of modular skilled birth attendant training package | "1 year"
  The health workers who get new modular skill birth attendant training are expected to be more competent to provide midwifery services. Hence, this training is specifically targeted to improve midwifery knowledge, attitudes, and skills.

SECONDARY OUTCOMES:
Cost-benefit analysis | "2 years"
  The associated cost (monetary value) of the new modular and standard training will be calculated and compared with the effect (maternal and neonatal death reduction).

CONTACTS AND LOCATIONS:
Overall Officials: Khim Bahadur Khadka, MPH, Principal Investigator — MoHP, HD, Gandaki
Locations (2):
- Nepal (2):
  - Health Directorate, Pokhara, Gandaki
  - Khim Bahadur Khadka, Pokhara, Gandaki

IPD SHARING:
Plan to Share IPD: No